CLINICAL TRIAL: NCT01454921
Title: A Secondary Prevention Empowerment Intervention for Young Women Living With HIV
Brief Title: Development of an Empowerment Intervention for Young Women Living With HIV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ATN 089
Record Dates: First submitted 2010-08-31; First posted 2011-10-19 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2016-03

CONDITIONS: HIV
Keywords: HIV; Adolescent Trials Network

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention I (Experimental): Intervention group participants will be enrolled for the duration of one intervention program, which will last approximately 6 months. Each intervention program will consist of two individual and six group intervention sessions with each session lasting approximately 2-3 hours.
  Intervention participants will also complete two ACASI assessments (baseline and post-intervention) lasting approximately 1.5-2 hours each.
  Interventions: Behavioral: Evolution: Young Women Taking Charge and Growing Stronger
- Intervention II (Experimental): Intervention group participants will be enrolled for the duration of one intervention program, which will last approximately 6 months. Each intervention program will consist of two individual and six group intervention sessions with each session lasting approximately 2-3 hours.
  Intervention participants will also complete two ACASI assessments (baseline and post-intervention) lasting approximately 1.5-2 hours each.
  Interventions: Behavioral: Evolution: Young Women Taking Charge and Growing Stronger

INTERVENTIONS:
Behavioral: Evolution: Young Women Taking Charge and Growing Stronger — The intervention aims to address the following concerns: 1) reducing the risk of young women infected with HIV transmitting the virus to their sexual partners, and 2) preventing young women infected with HIV from re-infection with a new viral strain or co-infection with another sexually transmitted disease (STD).

SUMMARY:
This study will develop/adapt a culturally appropriate secondary prevention intervention for young, Human Immunodeficiency Virus (HIV)-positive women through intervention groups, evaluate its acceptability and feasibility, make appropriate modifications, and manualize the intervention in preparation for a full-scale randomized trial.

Once the intervention is developed/adapted, the sites will pilot the interventions twice to enable modifications. The intervention aims to address the following concerns: 1) reducing the risk of young women infected with HIV transmitting the virus to their sexual partners, and 2) preventing young women infected with HIV from re-infection with a new viral strain or co-infection with another sexually transmitted disease (STD). Data will be collected to assess the feasibility and acceptability of the newly developed intervention using both quantitative and qualitative methods at each iteration.

ELIGIBILITY:
Inclusion Criteria:

* Female at birth and currently female;
* Receives services at one of the selected ATN sites or their community partners
* HIV-infected as documented by medical record review or verbal verification with referring professional
* Between the ages of 16-24 years (inclusive) at the time of informed consent/assent
* Ability to understand both written and spoken English
* Gives informed consent/assent for study participation

Exclusion Criteria:

* Presence of active, serious psychiatric symptoms (e.g., hallucinations, thought disorder) that would impair a participant's ability to meet the study requirements
* Visibly distraught (e.g., suicidal, homicidal, exhibiting violent behavior)
* Intoxicated or under the influence of alcohol or other substances at the time of study enrollment*.

  * Intoxication at the time of visit will exclude participation at that time. Participants cannot be visibly under the influence of substances at the time of enrollment or consent. If a participant returns to enroll while sober, enrollment can occur. Similarly, if a participant arrives to an intervention group visibly intoxicated, then she will be asked to leave. However, prior intoxication does not eliminate future participation. Thus, those who are dismissed from a session due to intoxication can return to a subsequent session as long as they are sober.

Ages: 16 Years to 24 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 43 (Actual)
Dates: Start 2010-02; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Compare pre-intervention, immediate post-intervention, and 3-month post-intervention scores on sexual risk and psychological empowerment | 1 year
  Compare pre-intervention ACASI scores on Sexual Activity and Sexual Risk and Psychological Empowerment Questionnaires with those collected immediately post-intervention and 3 months after intervention to determine effect of intervention on sexual risk and psychological empowerment.

SECONDARY OUTCOMES:
Compare pre-intervention, immediate post-intervention, and 3-month post-intervention scores on self-efficacy, sexual negotiation, relational violence, forgiveness, anger, substance use, life goals and outcomes, and affect regulation | 1 year
  Compare pre-intervention ACASI scores on three self-efficacy scales, two sexual negotiation scales, the Rosenberg Self-Esteem Scale, the CTS2, the HFS, the TAS, the ASSIST, a life goals/outcomes scale, and the Affect Regulation Scale with those collected immediately post-intervention and 3 months after intervention to determine effect of intervention on sexual risk and psychological empowerment.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Zimet, PhD, Study Chair — Adolescent Trials Network
Locations (3):
- United States (3):
  - USF College of Medicine, Tampa, Florida
  - Ruth M Rothstein CORE Center/ John H Stroger Jr Hospital, Chicago, Illinois
  - University of Maryland Medical School, Baltimore, Maryland

REFERENCES:
- See also: ATN Website — http://www.atnonline.org